CLINICAL TRIAL: NCT01398202
Title: Comparison of the Bioefficacy of Oral 25-hydroxyvitamin D3 and Vitamin D3 Supplements on Vitamin D Status in Older Adults
Brief Title: Dietary Supplementation With 25-hydroxyvitamin D3 in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Kevin D. Cashman, Professor of Food and Health, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 111
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Vitamin D Status as Reflected by Serum 25-hydroxyvitamin D
Keywords: Vitamin D status; 25-hydroxyvitamin D; Vitamin D3; RCT; Bio-efficacy
MeSH Terms: interventions — Cholecalciferol; Calcifediol; 25-hydroxyvitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D3 (20 microgram/day) (Active Comparator)
  Interventions: Dietary Supplement: vitamin D3
- 25-hydroxyvitamin D (7 microgram/day) (Active Comparator)
  Interventions: Dietary Supplement: 25-hydroxyvitamin D3
- 25-hydroxyvitamin D3 (20 micogram/day) (Active Comparator)
  Interventions: Dietary Supplement: 25-hydroxyvitamin D (20 microgram/day)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D3 — 20 micrograms per day for 10 weeks
  Arms: Vitamin D3 (20 microgram/day)
Dietary Supplement: 25-hydroxyvitamin D3 — 7 microgram/day for 10 weeks
  Arms: 25-hydroxyvitamin D (7 microgram/day)
Dietary Supplement: 25-hydroxyvitamin D (20 microgram/day) — 20 microgramday for 10 weeks
  Arms: 25-hydroxyvitamin D3 (20 micogram/day)
Dietary Supplement: Placebo — 0 ug vitamin D3/25-hydroxyvitamin D3/day for 10 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether a supplement of 25-hydroxyvitamin D is five-times more potent in raising vitamin D status (as reflected by serum 25(OH)D) compared to an equivalent amount of vitamin D3 in older adults. It will entail a 10 week supplementation study during winter months.

DETAILED DESCRIPTION:
The UK (McCance & Widdowson) food composition tables suggests that 25-hydroxyvitamin D (which is present in some foods, albeit at very low concentrations, but which is also commercially available) may possess up to 5-times the activity of native vitamin D3 in food. Thus, in theory, each micogram of 25-hydroxyvitamin D consumed in the diet could boost vitamin D status up to five times most effectively compared to each microgram of native vitamin D in food. It is worth noting, however, that estimates of potency range from 2 to 5, depending on approach used, and that the real potency needs to be confirmed in a human study. This study aims to examine the biological activity of 25-hydroxyvitamin D (i.e., its potency relative to vitamin D3) as well as its effect on selected functional markers in a randomised, double-blind, human intervention trial in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if they are 45+ years of age
* Body Mass Index (BMI) 19-30

Exclusion Criteria:

* have hypercalcaemia
* chronic illness
* renal or liver disorders
* taking medications that might interact with vitamin D or metabolite
* drank more than > 21 standards (male)/ 14 standards (female) of alcohol per week
* planning to change smoking habits

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
serum 25-hydroxyvitamin D concentration | 10 weeks

SECONDARY OUTCOMES:
serum parathyroid hormone | 10 weeks
blood pressure | 10 weeks
biochemical markers of bone turnover | 10 weeks
serum calcium adjusted for albumin | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Cashman, PhD, Principal Investigator — University College Cork
Locations (1):
- University College Cork, Cork, Ireland

REFERENCES:
- [Derived] Cashman KD, Seamans KM, Lucey AJ, Stocklin E, Weber P, Kiely M, Hill TR. Relative effectiveness of oral 25-hydroxyvitamin D3 and vitamin D3 in raising wintertime serum 25-hydroxyvitamin D in older adults. Am J Clin Nutr. 2012 Jun;95(6):1350-6. doi: 10.3945/ajcn.111.031427. Epub 2012 May 2. PMID 22552038